CLINICAL TRIAL: NCT02852603
Title: Study on Genetically Affected Sporadic Thoracic Aortic Aneurysm and Dissection
Acronym: GenSTAND
Status: Completed | Type: Observational
Sponsor: Wuhan Asia Heart Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Xuan Zheng, vice director of laboratory of molecular cardiology, Wuhan Asia Heart Hospital
Other Study IDs: 2016LMC-2
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Dissection of Aorta, Thoracic; Aneurysm of Aorta, Thoracic
Keywords: dissection; aneurysm; thoracic aorta
MeSH Terms: conditions — Aortic Dissection; Aortic Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral whole blood is obtained from patients. Serum, blood cell and DNA are separated and stored for further study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- thoracic aortic aneurysm and dissection: Patients with thoracic aortic aneurysm and/or dissection are recruited in the study.

SUMMARY:
Mortality of thoracic aortic aneurysm and dissection (TAAD) remains high because of the huge blood lost from the aorta. Questions about the potentially genetic effects on sporadic TAAD are raised by researchers to explore the possible mechanisms leading to sporadic TAAD and to establish new clinical approaches to prevent TAAD-caused adverse clinical outcomes. This study is intended to collect the gene information in sporadic TAAD patients and to explore the relationship between genetic variation and the incidence of sporadic TAAD for further study.

DETAILED DESCRIPTION:
Thoracic aortic dissection (TAD) is a critical clinical condition partly due to the rupture of aortic aneurysm. Mostly, surgical treatment can reduce the symptoms and extend life span of patients with thoracic aortic aneurysm and dissection (TAAD). However, mortality of TAAD remains high because of the huge blood lost from the aorta. Sporadic TAAD was considered to be a server consequence of hypertension, though most patients with hypertension won't have TAAD as their final outcomes. Previous studies have revealed the associations between genetic abnormalities and familial TAAD, and genetic tests have applied to assist the diagnosis of certain TAAD. Therefore, the potentially genetic effects on sporadic TAAD are explored by researchers to understand the possible mechanisms leading to sporadic TAAD and to establish new clinical approaches to prevent TAAD-caused adverse clinical outcomes. This study is intended to collect the gene information in sporadic TAAD patients and to explore the relationship between genetic variation and the incidence of sporadic TAAD for further study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thoracic aortic aneurysm and dissection not due to trauma

Exclusion Criteria:

* Inability of the patient, parent or guardian to give consent
* Unwillingness to provide a blood specimen or participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thoracic aortic aneurysm and dissection.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Numbers of patients having thoracic aortic aneurysm and/or dissection are recorded. Diagnosis are confirmed by imaging analysis (CTA and/or Ultrasound) or by doctors during the operations. | 6 months
  Arterial dissection actually happened

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zheng, MD, PhD, Principal Investigator — Wuhan Asia Heart Hospital
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided